CLINICAL TRIAL: NCT03504319
Title: The Role of Physical Activity During Pregnancy on Metabolic Function, Inflammation, and Maternal and Neonatal Outcomes
Status: Completed | Type: Observational
Sponsor: Western Kentucky University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-229; 5P20GM1034 (Other Grant/Funding Number: NIH NIGMS IDeA Grant)
Record Dates: First submitted 2018-03-29; First posted 2018-04-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Obesity; Pregnancy Related
Keywords: exercise; inflammation; metabolic inflexibility; insulin resistance; neonatal adiposity
MeSH Terms: conditions — Obesity; Motor Activity; Inflammation; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — maternal- whole blood, red blood cells (after spinning and removing plasma), plasma cord blood- cord blood plasma, cord blood red blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lean Group: Pre-pregnancy BMI between 18.5 and 24.9 kg/m2
  Interventions: Other: Exposure to high-fat smoothie
- Obese Group: Pre-pregnancy BMI ≥30 kg/m2
  Interventions: Other: Exposure to high-fat smoothie

INTERVENTIONS:
Other: Exposure to high-fat smoothie — Both groups will drink the high-fat smoothie and the study team will observe how they respond metabolically in the subsequent four hours using metabolic analyzer and blood draws.

SUMMARY:
Maternal obesity during pregnancy is a serious public health concern as it contributes to inflammation, insulin resistance, and excessive gestational weight gain- all of which negatively impact maternal and neonatal health. Fortunately, physical activity during pregnancy improves obstetric and infant outcomes associated with obesity. Specifically, data from our group demonstrated that irrespective of body weight, women who were physically-active during pregnancy had lower levels of systemic inflammation; however, the mechanism/s driving these changes are poorly understood. Previous studies in non-gravid populations suggest obesity-associated overnutrition may contribute to inflammation and this subsequent inflammation may lead to further metabolic dysfunction- perpetuating a vicious cycle. However, the connections between physical activity, inflammation, and metabolic dysfunction (i.e. metabolic inflexibility), particularly in response to a high-fat meal (similar to that which is typically consumed in a Western diet), among lean and obese pregnant women have not been studied. Thus, this study will examine the impact of a physically-active lifestyle on inflammatory and metabolic responses to a high-fat meal in lean and obese pregnant women. Understanding mechanisms connecting maternal physical activity to improved outcomes will better inform future targeted intervention strategies. The goal of this study is to determine the role of a physically-active lifestyle during pregnancy on metabolic function and inflammation following a high-fat meal in lean and obese pregnant women.

DETAILED DESCRIPTION:
Maternal obesity is a significant public health concern in the United States as one in three women enter pregnancy obese, and maternal obesity is associated with a large number of unfavorable maternal and neonatal outcomes. Fortunately, a physically active lifestyle during pregnancy has been shown to improve unfavorable outcomes often associated with obesity. Physical activity during pregnancy has been shown to improve maternal insulin resistance and reduce maternal gestational weight gain. In addition, neonates of physically active women have lower adiposity compared to neonates born to inactive women. Although the relationships between physical activity and maternal and neonatal outcomes are well-established, little is known about the potential for metabolic dysfunction and/or inflammation to serve as mechanisms mediating the positive impact of physical inactivity on maternal and neonatal health. Understanding mechanisms connecting maternal physical activity to improved outcomes will better inform future targeted intervention strategies.

Metabolic adaptations, specifically changes in lipid and carbohydrate metabolism, occur during normal physiologic pregnancy to provide an adequate nutrient supply to the developing fetus despite intermittent maternal dietary intake. However, in obese pregnant women these metabolic adaptations may be augmented by additional maternal metabolic dysfunction. Further, it is well-established that metabolic dysfunction in obese pregnant women has serious implications for maternal and neonatal health. Maternal substrate metabolism not only contributes to maternal health conditions such as gestational diabetes, but it also plays a major role in fetal growth and development. The "fetal origins hypothesis" suggests that an altered intrauterine metabolic environment may contribute to the programming of short and long-term neonatal outcomes.

Metabolic inflexibility may play a major role in maternal and neonatal health; however, it has not been studied during pregnancy. In non-gravid populations, physical activity is positively correlated with metabolic flexibility, and physical activity improves metabolic flexibility in lean and obese individuals.

The role of physical activity in modulating metabolic inflexibility in lean and obese pregnant women has not been studied. However, an impaired ability to switch to fat metabolism after a high-fat load is likely a better indicator of metabolic dysregulation than metabolism during resting conditions. Therefore, the current study proposes to look at the role of a physically active lifestyle on metabolic function in lean and obese pregnant women.

This project will also determine the relationships between inflammation, metabolic flexibility, and other important maternal (gestational weight gain) and neonatal (adiposity and insulin resistance) outcomes.The goal of this project is to investigate the impact of a physically-active lifestyle on inflammatory and metabolic responses to a high-fat meal in lean and obese pregnant women.

The investigators hypothesize that a physically-active lifestyle among lean and obese pregnant women will improve metabolic function and inflammation thus mediating the positive effects of physical activity on maternal and neonatal health outcomes

Sixty women (30 lean, 30 obese) will be recruited between 28-32 weeks of pregnancy.

Consent and Physical Activity Assessment The study team will meet and consent the patient at a private office. Participants will be given an Actigraph Link Accelerometer (ActiGraph LLC, Pensacola, FL) to objectively confirm their self-reported physical activity levels. The Link will be placed on the non-dominant wrist with non-removable hospital-grade wristbands. Wrist-worn tri-axel accelerometers are a valid measure of physical activity energy expenditure in pregnant women. In addition, previous data on acceptability suggest participants do not object to wearing wrist-worn devices 24 hours/day, and we believe wrist-worn devices with hospital-type wristbands would give us the best compliance and 24 hours/day wear data. Data will be collected for seven consecutive days at 30 Hz. The accelerometer output will be sampled by a 12-bit analog-to-digital converter. The percentage of time spent sedentary as well as the amount of time spent participating in different categories of physical activity ranging from light and lifestyle to moderate will be calculated using algorithms corresponding to the following activity counts: sedentary: 0 - 99 counts/min, light: 100 - 759 counts/min, lifestyle: 760 - 1951 counts/min, moderate: 1952-5724 counts/min.

Maternal Metabolic Inflexibility and Inflammation in Response to a High-Fat Meal Participants will report to the Exercise Laboratory located on the Medical Health Complex in Bowling Green, KY at approximately 8:00am after a 10-hour fast. Participants will be provided with written instructions for consuming a standardized diet the day before with approximately 50% carbohydrate, 30% fat, and 20% protein. The participant's weight, height, and vitals will be taken upon arrival. Body composition will be measured using skinfold anthropometry in order to determine maternal percent body fat. Body fat percentage will be determined by pressing folds of the skin at seven sites with a caliper (Harpenden Skinfolds Caliper, Baty International, United Kingdom), recording skin fold thickness, and entering the data into a standardized equation that accounts for age, a technique that has been used during pregnancy in prior studies.

Resting metabolic rate and respiratory quotient will be measured for ~30minutes using the TrueOne Canopy Option and TrueOne Metabolic Cart (TrueOne 2400, Parvomedics, Sandy, UT). Lipid and carbohydrate oxidation rates will be calculated by measurement of oxygen consumption and carbon dioxide production as previously described. After the baseline resting metabolism measurement, a baseline blood draw will be obtained (time point- 0). After the baseline blood draw, participants will consume a standard 1000-kcal meal that is high in fat, similar in composition to previous studies. The high-fat meal will consist of a Smoothie from Smoothie King (55.9% fat, 29.4% carbs, 14.7% protein). Additional blood samples will be taken 60, 120, and 240 minutes after the meal is consumed. Resting metabolic rate and respiratory quotient will be obtained a second time for ~30minutes from minute 210 to 240 minutes post meal consumption. A total of 32mL maternal blood will be drawn. Time points for assessment of metabolic responses to a high-fat load were chosen based on data from previous studies exploring metabolic inflexibility and inflammation in response to a high-fat meal in other populations.

Blood draws will be used to analyze maternal plasma glucose, insulin, c-peptide, free fatty acids, lipids (triglycerides, HDL, LDL), and inflammatory markers (IL-6, TNF-α, IL-1α). All blood samples will be analyzed using standardized protocols at the Biochemistry Lab at WKU or the Washington University Core Laboratory for Clinical Studies. These data will provide additional information regarding metabolic responses to the high-fat load. Baseline insulin and glucose levels will be used to calculate the homeostatic model assessment-insulin resistance (HOMA-IR), an index of insulin resistance that reflects fasting glucose concentration measured at the fasting insulin concentration. Data on each participants' oral glucose tolerance test (performed ~24-28 weeks gestation) will also be obtained from prenatal charts to examine insulin resistance.

During the four hour study period, participants will be asked to remain reclined and resting. Participants will complete several surveys during this time as well including the National Institutes of Health's validated Dietary History Questionnaire II to determine potential differences in day-to-day diet and the Pregnancy Physical Activity Questionnaire to determine domain and mode of physical activities.

Neonatal Outcomes At parturition, neonatal weight, length, and head circumference will be obtained via labor and delivery nurses. Approximately 20mL umbilical cord blood will be obtained, centrifuged within one hour of delivery, and placed in a -80º C freezer. Neonatal insulin, glucose, inflammatory markers (IL-6, TNF-α, IL-1α), and free fatty acids will be determined from the umbilical cord plasma.

Within 48 hours of delivery, neonatal body composition (fat and lean mass) will be measured by skin fold thickness measurement at the patients' bedside. Maternal prenatal charts will be obtained in order to determine gestational weight gain and any other medical conditions that may influence the interpretation of study outcomes.

Statistical Procedures Sample Size Calculation Due to the lack of data regarding metabolic inflexibility during pregnancy and the exploratory nature of the study, data from a previous study comparing metabolic inflexibility between several non-gravid populations using the same methodology as the current study was used, where 29 subjects per group would provide 80% power to detect differences in metabolic flexibility (via indirect calorimetry) between active and inactive pregnant women.

Statistical Analyses Normality of the distribution for each variable will be tested using Kolmogorov-Smirnov tests. Pearson product-moment correlation coefficients for normally distributed variables or Spearman's rank-order correlation coefficient for non-normally distributed variables will be used to assess the degree of the relationship between variables. Partial correlations will be used to adjust for potential confounders. Student's independent t-tests for normally distributed variables and Mann-Whitney U tests for non-normally distributed variables will be used to compare outcomes between lean and obese pregnant women. All tests will be two-sided with a p-value <0.05 denoting statistical significance. All data analyses will be conducted using IBM SPSS Statistics, Version 22 (Armonk, New York).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-44
* Confirmed singleton viable pregnancy with no fetal abnormalities at routine 18-22 ultrasonography
* Receipt of prenatal care and plans to deliver at The Medical Center in Bowling Green, KY
* Completion of a normal routine, standard of care gestational diabetes screen
* Physician release to participate in the study procedures

Exclusion Criteria:

* Multiple gestation pregnancy
* Inability to provide voluntary informed consent
* Current use of illegal drugs (cocaine, methamphetamine, opiates, etc…)
* Current smoker who does not consent to cessation
* Current usage of daily medications by class: corticosteroids, anti-psychotics (known to alter insulin resistance and metabolic profiles)
* History of gestational diabetes, pre-pregnancy diabetes or prior macrosomic (>4500g) infant (each elevate the risk for gestational diabetes in the current pregnancy, or undiagnosed gestational diabetes)
* Dietary restrictions prohibiting them from consuming the standardized meal/high-fat load

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from several local obstetrics offices, as well as through word of mouth, university-wide emails, and local flyers (with IRB approval).
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in metabolic inflexibility | Metabolic inflexibility will be assessed 2 and 4 hours after shake consumption
  The increase in fat metabolism after smoothie consumption (lipid oxidation in g/min after shake minus lipid oxidation (g/min) before shake/ lipid oxidation before shake (g/min))

SECONDARY OUTCOMES:
Change in inflammation | Inflammatory markers will be assessed at baseline, 2 hours, and 4 hours post smoothie consumption
  Markers of inflammation (assessed via pro-inflammatory cytokines for IL-6, IL-alpha, TNF-alpha, CRP)
Maternal gestational weight gain | Maternal weight at delivery will be obtained from her last reported weight before delivery, pre-pregnancy weight will be determined from self-report at study enrollment (~28 weeks)
  Maternal weight at delivery (kg) minus maternal pre-pregnancy weight (kg)
Neonatal insulin | At delivery
  From cord blood plasma (μU/ml)
Neonatal glucose | At delivery
  From cord blood plasma (mmol/L)
Neonatal insulin resistance | At delivery
  Homeostatic Model Assessment- Insulin Resistance ((neonatal insulin x neonatal glucose)/405)
Change in maternal insulin | At baseline, 2 hours, and 4 hours post shake consumption
  From maternal plasma (μU/ml)
Change in maternal glucose | At baseline, 2 hours, and 4 hours post shake consumption
  From maternal plasma (mmol/L)
Change in maternal insulin resistance | At baseline, 2 hours, and 4 hours post shake consumption
  Insulin resistance will be assessed via a homeostatic assessment of insulin resistance (HOMA-IR) using glucose and insulin concentrations from maternal blood ((glucose x insulin)/405)
Neonatal adiposity | 24-48 hours post delivery
  Peapod air displacement plethysmography (% body fat)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Tinius, PhD, Principal Investigator — Western Kentucky University
Locations (1):
- Western Kentucky University, Bowling Green, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided